CLINICAL TRIAL: NCT04223349
Title: A Phase 1, Open-label Single-dose Crossover, and Double-blind Multiple-dose Parallel Group Study to Characterize the Pharmacokinetics, Safety and Tolerability, and Pharmacodynamics of JNJ-70033093 in Healthy Adult Subjects
Brief Title: A Study of JNJ-70033093 (BMS-986177) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR108728; 70033093THR1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-01-08; First posted 2020-01-10 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — milvexian

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part 1: Treatment A (Experimental): Participants will receive JNJ-70033093 dose twice daily (BID) for 8 days followed by a placebo dose on Day 9 or placebo BID for 8 days followed by a placebo dose on Day 9.
  Interventions: Drug: JNJ-70033093; Drug: Placebo
- Part 1: Treatment B (Experimental): Participants will receive JNJ-70033093 dose BID for 8 days followed by a placebo dose on Day 9 or placebo BID for 8 days followed by a placebo dose on Day 9.
  Interventions: Drug: JNJ-70033093; Drug: Placebo
- Part 1: Treatment C (Experimental): Participants will receive JNJ-70033093 dose BID for 8 days followed by a JNJ-70033093 dose on Day 9 or placebo BID for 8 days followed by a placebo dose on Day 9.
  Interventions: Drug: JNJ-70033093; Drug: Placebo
- Part 1: Treatment D (Experimental): Participants will receive JNJ-70033093 dose BID for 8 days followed by a JNJ-70033093 dose on Day 9 or placebo BID for 8 days followed by a placebo dose on Day 9.
  Interventions: Drug: JNJ-70033093; Drug: Placebo
- Part 2: Treatment Sequence EFG (Experimental): Participants will receive Treatment E (JNJ-7003309 single dose in the morning in fasted condition) in treatment Period 1; followed by Treatment F (JNJ-7003309 single dose administered in the evening in fasted condition) in treatment Period 2; followed by Treatment G (JNJ-7003309 single dose administered in the evening in fasted condition) in treatment Period 3, on Day 1 of each treatment period. A washout period of at least 4 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-70033093
- Part 2: Treatment Sequence FGE (Experimental): Participants will receive Treatment F in treatment Period 1; followed by Treatment G in treatment Period 2; followed by Treatment E in treatment Period 3, on Day 1 of each treatment period. A washout period of at least 4 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-70033093
- Part 2: Treatment Sequence GEF (Experimental): Participants will receive Treatment G in treatment Period 1; followed by Treatment E in treatment Period 2; followed by Treatment F in treatment Period 3, on Day 1 of each treatment period. A washout period of at least 4 days will be maintained between each treatment period
  Interventions: Drug: JNJ-70033093
- Part 2: Treatment Sequence EGF (Experimental): Participants will receive Treatment E in treatment Period 1; followed by Treatment G in treatment Period 2; followed by Treatment F in treatment Period 3, on Day 1 of each treatment period. A washout period of at least 4 days will be maintained between each treatment period
  Interventions: Drug: JNJ-70033093
- Part 2: Treatment Sequence GFE (Experimental): Participants will receive Treatment G in treatment Period 1; followed by Treatment F in treatment Period 2; followed by Treatment E in treatment Period 3, on Day 1 of each treatment period. A washout period of at least 4 days will be maintained between each treatment period
  Interventions: Drug: JNJ-70033093
- Part 2: Treatment Sequence FEG (Experimental): Participants will receive Treatment F in treatment Period 1; followed by Treatment E in treatment Period 2; followed by Treatment G in treatment Period 3, on Day 1 of each treatment period. A washout period of at least 4 days will be maintained between each treatment period
  Interventions: Drug: JNJ-70033093

INTERVENTIONS:
Drug: JNJ-70033093 — JNJ-70033093 capsules will be administered orally .
Drug: Placebo — Matching placebo in capsule will be administered orally.
  Arms: Part 1: Treatment A; Part 1: Treatment B; Part 1: Treatment C; Part 1: Treatment D

SUMMARY:
The purpose of this study is to characterize the pharmacokinetic (PK) of multiple twice-daily doses of JNJ-70033093 in healthy participants and to assess the effects of dosing time and food on the PK of single-dose of JNJ-70033093 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history, physical examination, vital signs, electrocardiogram (ECG), and laboratory test results, including serum chemistry, blood coagulation, hematology, and urinalysis performed at screening. If there are abnormalities, the investigator may decide that the abnormalities or deviations from normal are not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* If a woman, except for postmenopausal women, must have a negative highly sensitive serum (beta human chorionic gonadotropin [beta-hCG]) at screening and urine (beta-hCG) pregnancy test on Day -1 of treatment period
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participant participating in clinical studies
* Body mass index (BMI; weight kilogram per meter square [kg/m^2]) between 18 and 30 kg/m^2 (inclusive), and body weight not less than 50 kilogram (kg)
* After being supine for 10 minutes, systolic blood pressure between 90 and 140 millimeter of Mercury (mmHg), inclusive; and no higher than 90 mmHg diastolic blood pressure

Exclusion Criteria:

* If a woman, pregnant, breast-feeding or planning to become pregnant during the study
* History of any known illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant or that could prevent, limit or confound the protocol specified assessments. This may include but is not limited to any known bleeding or clotting disorder, a history of arterial or venous thrombosis, liver or renal dysfunction, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic abnormalities, metabolic disturbances, or poor venous access
* Participants with current hepatitis B infection (confirmed by hepatitis B surface antigen [HBsAg]), or hepatitis C infection (confirmed by hepatitis C virus [HCV] antibody), or human immunodeficiency virus type-1 (HIV-1) or HIV-2 infection at study screening
* History of, or a reason to believe a participant has a history of, drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM V) criteria within the past 1 year, which in the investigator's opinion would compromise participant safety and/or compliance with the study procedures
* History of any clinically significant drug or food allergies (such as anaphylaxis or hepatotoxicity) and known allergy to the study drugs or any of the excipients of the formulation. History of allergy to or unwillingness to consume any component of the high-fat breakfast menu to be provided in this study
* Clinically significant abnormal values for hematology, coagulation, clinical chemistry or urinalysis at Screening or on Day -1 prior to the first dosing as determined by the investigator or appropriate designee. Any of the following laboratory results outside of the ranges specified below at screening or Day -1 prior to first dosing, confirmed by repeat: Hemoglobin or hematocrit < lower limit of normal; Platelet count < lower limit of normal; activated partial thromboplastin time (aPTT), or prothrombin time (PT) greater than (>) 1.2 × upper limit of normal (ULN)
* Any of the following on 12-lead ECG and assessment of QT interval prior to study treatment administration, confirmed by repeat at screening and Day -1 of treatment period: Heart rate >100 beats per minute (bpm); PR >= 210 milli second (ms); QRS >=120 ms; QTcF >= 450 ms for male and >= 470 ms for female

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum Observed Analyte Concentration (Cmax) of JNJ-70033093 | Up to Day 9
  Cmax is the maximum observed analyte concentration.
Part 1: Time to Reach the Maximum Observed Analyte Concentration (Tmax) of JNJ-70033093 | Up to Day 9
  Tmax is the actual sampling time to reach the maximum observed analyte concentration
Part 1: Area Under the Analyte Concentration-time Curve from Time Zero to 12 Hours (AUC[0-12h]) of JNJ-70033093 | 12 hours postdose (Day 1)
  AUC(0-12h) is the area under the time-concentration curve (AUC) from time 0 (dosing time) to 12 hours before steady state.
Part 1: Apparent Terminal Elimination Half-life (t[1/2]) of JNJ-70033093 | Up to Day 9
  T(1/2) is the apparent terminal elimination half-life is the time measured for the analyte concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Part 2: Maximum Observed Analyte Concentration (Cmax) of JNJ-70033093 | Up to Day 9
  Cmax is the maximum observed analyte concentration.
Part 2: Area Under the Concentration-time Curve from Time Zero to the Last Measurable Concentration (AUC [0-last]) of JNJ-70033093 | Up to Day 9
  AUC (0-last) is area under the analyte concentration-time curve (AUC) from time 0 to time of the last quantifiable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Part 2: Area Under the Concentration-time Curve from Time Zero to Infinity (AUC [0-infinity]) of JNJ-70033093 | Up to Day 9
  AUC (0-infinity) is the area under the analyte concentration-time curve (AUC) from time zero to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration-time curve from time zero to last measurable concentration, C(last) is the last observed measurable (non-BQL) analyte concentration; and lambda(z) is apparent terminal elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 51 days
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product does not necessarily have a causal relationship with the treatment.
Number of Participants with Vital Sign Abnormalities | Up to 51 days
  Number of participants with vital signs (including body temperature, resting [supine] pulse rate, and blood pressure) abnormalities will be reported.
Number of Participants with Abnormal Electrocardiogram (ECG) Findings | Up to 51 days
  Number of participants with abnormal ECG findings will be reported.
Number of Participants with Abnormal Laboratory Findings | Up to 51 days
  Number of participants with abnormal laboratory findings (that is, hematology, coagulation tests, clinical chemistry, urinalysis) will be reported.
Relationship Between JNJ-70033093 Plasma Concentrations and QTc After Multiple Doses of JNJ-70033093 | Up to Day 9
  Relationship between JNJ-70033093 plasma concentrations and QTc in healthy participants receiving multiple doses of JNJ-70033093 will be assessed.
Percentage Change from Baseline in Activated Partial Thromboplastin Time (aPTT) | Baseline up to Day 9 (Part 1); Baseline up to Day 11 (Part 2)
  aPTT measures the time to clot formation via the contact and common activation pathway. Blood will be collected for measurement of changes in aPTT clotting time.
Percentage Change from Baseline in Factor XI Clotting Activity | Baseline up to Day 9 (Part 1); Baseline up to Day 11 (Part 2)
  Percentage change from baseline in FXI clotting activity will be measured using a modified aPTT assay.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency